CLINICAL TRIAL: NCT00468923
Title: Heart Outcomes Prevention Evaluation-3
Acronym: HOPE-3
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Responsible Party: Principal Investigator, Salim Yusuf's office, Principal Investigator, Population Health Research Institute
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HOPE-3
Record Dates: First submitted 2007-05-02; First posted 2007-05-03 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Cardiovascular Disease; Stroke
Keywords: Primary prevention; Cholesterol lowering; Blood pressure lowering; Cardiovascular disease prevention
MeSH Terms: conditions — Cardiovascular Diseases; Stroke | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rosuvastatin (Placebo Comparator): Rosuvastatin 10 mg vs placebo
  Interventions: Drug: Rosuvastatin
- Candesartan/HCT (Placebo Comparator): Candesartan 16 mg/HCT 12.5 mg vs placebo
  Interventions: Drug: Candesartan/HCT

INTERVENTIONS:
Drug: Candesartan/HCT — Candesartan 16 mg/HCT 12.5 once daily
  Arms: Candesartan/HCT
Drug: Rosuvastatin — Rosuvastatin 10 mg once daily
  Arms: Rosuvastatin

SUMMARY:
Heart disease and stroke are major causes of death and disability worldwide and are largely preventable. Cholesterol and blood pressure are major cardiovascular risk factors. Previous studies have shown that certain drugs can effectively and safely lower cholesterol and blood pressure and prevent heart attacks and strokes. Such studies have been conducted primarily in people who had already sustained a heart attack or a stroke, or in people with high cholesterol and blood pressure levels. However, most heart attacks and strokes occur in people with average ("normal") cholesterol and blood pressure. Therefore, in the HOPE-3 trial the investigators will evaluate whether a cholesterol lowering drug, rosuvastatin, and a combination blood pressure lowering pill, candesartan/hydrochlorothiazide, used alone or together can reduce the risk of heart attacks, stroke and their sequelae in people without known heart disease and at average risk.

DETAILED DESCRIPTION:
The trial has randomized 12,705 women 60 years or older and men 55 years or older without known heart disease or prior stroke and without a clear indication or contraindication to any of the study medications. Eligible and consenting individuals were randomized to receive either active study medications or placebo (dummy pills) and will be monitored for an average of 5.7 years. The rates of heart attacks, strokes, deaths and other cardiovascular events will be compared between subjects receiving the active drugs and those on placebo. The study included people from 21 countries, which were monitored by an international group of scientists and physicians. The study was coordinated by the Population Health Research Institute at McMaster University. The study is expected to demonstrate that combined lipid lowering and blood pressure lowering will substantially lower the risk for cardiovascular diseases and may substantially change our approach to cardiovascular prevention.

ELIGIBILITY:
Inclusion Criteria:

* Women aged > 60 years and men > 55 years
* At least one additional CV risk factor including:
* Waist/hip ratio ≥ 0.90 in men and ≥ 0.85 in women;
* History of current or recent smoking (regular tobacco use within 5 years)
* Low HDL cholesterol
* Dysglycemia
* Renal dysfunction
* Family history of premature CHD in first degree relatives

Exclusion Criteria:

* Documented clinically manifest atherothrombotic CVD
* Clear indication or contraindication for statin and/or ARB or ACE inhibitor and/or thiazide diuretic therapy
* Symptomatic hypotension
* Chronic liver disease
* Inflammatory muscle disease
* Renal impairment
* Concurrent treatment with cyclosporine or a condition likely to result in organ transplantation and the need for cyclosporine
* Concurrent treatment with a statin, fibrate, angiotensin receptor blocker, ACE inhibitor, or a thiazide diuretic
* Other serious medical illness likely to interfere with study participation or with the ability to complete the trial
* Significant psychiatric illness, senility, dementia, alcohol or substance abuse, which could impair the ability to provide informed consent and to adhere to the trial procedures
* Concurrent use of an experimental pharmacological agent

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12705 (Actual)
Dates: Start 2007-05; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
The composite of; Cardiovascular death, non-fatal myocardial infarction, non-fatal stroke. | Biannually
The composite of; cardiovascular death, resuscitated cardiac arrest, non-fatal myocardial infarction, non-fatal stroke, heart failure, arterial revascularizations | Biannually

SECONDARY OUTCOMES:
Total mortality | Biannually
The components of the co-primary endpoints | Biannually

OTHER OUTCOMES:
Renal Dysfunction | Biannually
Arterial revascularizations. | Biannually
New diagnosis of diabetes. | Biannually
All components of the co-primary and secondary outcomes | Follow-up
Cognitive function | Follow-up
Erectile dysfunction in men | Biannually
Myopathy (defined as muscle aches or pains accompanied by CK rise >10ULN). | Biannually
Rhabdomyolysis (defined as muscle pain and/or weakness associated with CK rise >10 ULN and evidence of acute renal dysfunction). | Biannually
Hospital admissions and the reason for admission. | Biannually
Cancer | Biannually

CONTACTS AND LOCATIONS:
Overall Officials: Salim Yusuf, DPhil FRCPC, Principal Investigator — McMaster University; Eva Lonn, MD MSc FRCPC, Principal Investigator — McMaster University
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with participants in the study April/May 2016

REFERENCES:
- [Result] Lonn EM, Bosch J, Lopez-Jaramillo P, Zhu J, Liu L, Pais P, Diaz R, Xavier D, Sliwa K, Dans A, Avezum A, Piegas LS, Keltai K, Keltai M, Chazova I, Peters RJ, Held C, Yusoff K, Lewis BS, Jansky P, Parkhomenko A, Khunti K, Toff WD, Reid CM, Varigos J, Leiter LA, Molina DI, McKelvie R, Pogue J, Wilkinson J, Jung H, Dagenais G, Yusuf S; HOPE-3 Investigators. Blood-Pressure Lowering in Intermediate-Risk Persons without Cardiovascular Disease. N Engl J Med. 2016 May 26;374(21):2009-20. doi: 10.1056/NEJMoa1600175. Epub 2016 Apr 2. PMID 27041480
- [Result] Yusuf S, Bosch J, Dagenais G, Zhu J, Xavier D, Liu L, Pais P, Lopez-Jaramillo P, Leiter LA, Dans A, Avezum A, Piegas LS, Parkhomenko A, Keltai K, Keltai M, Sliwa K, Peters RJ, Held C, Chazova I, Yusoff K, Lewis BS, Jansky P, Khunti K, Toff WD, Reid CM, Varigos J, Sanchez-Vallejo G, McKelvie R, Pogue J, Jung H, Gao P, Diaz R, Lonn E; HOPE-3 Investigators. Cholesterol Lowering in Intermediate-Risk Persons without Cardiovascular Disease. N Engl J Med. 2016 May 26;374(21):2021-31. doi: 10.1056/NEJMoa1600176. Epub 2016 Apr 2. PMID 27040132
- [Result] Yusuf S, Lonn E, Pais P, Bosch J, Lopez-Jaramillo P, Zhu J, Xavier D, Avezum A, Leiter LA, Piegas LS, Parkhomenko A, Keltai M, Keltai K, Sliwa K, Chazova I, Peters RJ, Held C, Yusoff K, Lewis BS, Jansky P, Khunti K, Toff WD, Reid CM, Varigos J, Accini JL, McKelvie R, Pogue J, Jung H, Liu L, Diaz R, Dans A, Dagenais G; HOPE-3 Investigators. Blood-Pressure and Cholesterol Lowering in Persons without Cardiovascular Disease. N Engl J Med. 2016 May 26;374(21):2032-43. doi: 10.1056/NEJMoa1600177. Epub 2016 Apr 2. PMID 27039945
- [Derived] Dagenais GR, Pais P, Gao P, Roshandel G, Malekzadeh R, Joseph P, Yusuf S. Fixed dose combination therapies in primary cardiovascular disease prevention in different groups: an individual participant meta-analysis. Heart. 2023 Aug 24;109(18):1372-1379. doi: 10.1136/heartjnl-2022-322278. PMID 37258095
- [Derived] Bosch J, Lonn EM, Dagenais GR, Gao P, Lopez-Jaramillo P, Zhu J, Pais P, Avezum A, Sliwa K, Chazova IE, Peters RJG, Held C, Yusoff K, Lewis BS, Toff WD, Khunti K, Reid CM, Leiter LA, Yusuf S, Hart RG. Antihypertensives and Statin Therapy for Primary Stroke Prevention: A Secondary Analysis of the HOPE-3 Trial. Stroke. 2021 Aug;52(8):2494-2501. doi: 10.1161/STROKEAHA.120.030790. Epub 2021 May 14. PMID 33985364
- [Derived] Bosch J, Lonn EM, Jung H, Zhu J, Liu L, Lopez-Jaramillo P, Pais P, Xavier D, Diaz R, Dagenais G, Dans A, Avezum A, Piegas LS, Parkhomenko A, Keltai K, Keltai M, Sliwa K, Held C, Peters RJG, Lewis BS, Jansky P, Yusoff K, Khunti K, Toff WD, Reid CM, Varigos J, Joseph P, Leiter LA, Yusuf S. Lowering cholesterol, blood pressure, or both to prevent cardiovascular events: results of 8.7 years of follow-up of Heart Outcomes Evaluation Prevention (HOPE)-3 study participants. Eur Heart J. 2021 Aug 17;42(31):2995-3007. doi: 10.1093/eurheartj/ehab225. PMID 33963372
- [Derived] Khunti K, Jung H, Dans AL, Held C, Dagenais GR, Yusuf S, Lonn E. Statin Use in Primary Prevention: A Simple Trial-Based Approach Compared With Guideline-Recommended Risk Algorithms for Selection of Eligible Patients. Can J Cardiol. 2019 May;35(5):644-652. doi: 10.1016/j.cjca.2019.03.002. Epub 2019 Mar 19. PMID 31030865
- [Derived] Bosch J, O'Donnell M, Swaminathan B, Lonn EM, Sharma M, Dagenais G, Diaz R, Khunti K, Lewis BS, Avezum A, Held C, Keltai M, Reid C, Toff WD, Dans A, Leiter LA, Sliwa K, Lee SF, Pogue JM, Hart R, Yusuf S; HOPE-3 Investigators. Effects of blood pressure and lipid lowering on cognition: Results from the HOPE-3 study. Neurology. 2019 Mar 26;92(13):e1435-e1446. doi: 10.1212/WNL.0000000000007174. Epub 2019 Feb 27. PMID 30814321
- [Derived] Lamy A, Lonn E, Tong W, Swaminathan B, Jung H, Gafni A, Bosch J, Yusuf S. The cost implication of primary prevention in the HOPE 3 trial. Eur Heart J Qual Care Clin Outcomes. 2019 Jul 1;5(3):266-271. doi: 10.1093/ehjqcco/qcz001. PMID 30657891
- [Derived] Lonn E, Bosch J, Pogue J, Avezum A, Chazova I, Dans A, Diaz R, Fodor GJ, Held C, Jansky P, Keltai M, Keltai K, Kunti K, Kim JH, Leiter L, Lewis B, Liu L, Lopez-Jaramillo P, Pais P, Parkhomenko A, Peters RJ, Piegas LS, Reid CM, Sliwa K, Toff WD, Varigos J, Xavier D, Yusoff K, Zhu J, Dagenais G, Yusuf S; HOPE-3 Investigators. Novel Approaches in Primary Cardiovascular Disease Prevention: The HOPE-3 Trial Rationale, Design, and Participants' Baseline Characteristics. Can J Cardiol. 2016 Mar;32(3):311-8. doi: 10.1016/j.cjca.2015.07.001. Epub 2015 Jul 8. PMID 26481083